CLINICAL TRIAL: NCT04936542
Title: A Multicentre, Interventional, Post-marketing, Randomised, Double-blind, Crossover Study to Evaluate the Clinical Safety and Efficacy of AbobotulinumtoxinA (Dysport®) in Comparison With OnabotulinumtoxinA (Botox®) When Treating Adults With Upper Limb Spasticity
Brief Title: A Study to Compare the Safety and Efficacy of Dysport® and Botox® in Adults With Upper Limb Spasticity.
Acronym: DIRECTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-52120-452; 2021-000161-32 (EudraCT Number)
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Upper Limb Spasticity
MeSH Terms: interventions — abobotulinumtoxinA; onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): Participants will receive one cycle of aboBoNT-A followed by one cycle of onaBoNT-A in the selected overactive upper limb muscles
  Interventions: Biological: AboBoNT-A; Biological: OnaBoNT-A
- Sequence 2 (Other): Participants will receive one cycle of onaBoNT-A followed by one cycle of aboBoNT-A in the selected overactive upper limb muscles
  Interventions: Biological: AboBoNT-A; Biological: OnaBoNT-A

INTERVENTIONS:
Biological: AboBoNT-A — AbobotulinumtoxinA for injection: 500 Unit vial. Dose: 900 Units (3.6 mL)
  Other Names: Dysport®
Biological: OnaBoNT-A — OnabotulinumtoxinA for injection: 200 Unit vial. Dose: 360 Units (3.6 mL)
  Other Names: Botox®

SUMMARY:
This study is aiming to demonstrate the non-inferiority of AbobotulinumtoxinA (aboBoNT-A) versus OnabotulinumtoxinA (onaBoNT-A) as the primary safety endpoint, and the superiority of aboBoNT-A over onaBoNT-A with respect to duration of response as the key secondary efficacy endpoint when used at optimal doses according to approved prescribing information of each product.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent
* 2a. [US/France] Participants with stable Upper Limb Spasticity (ULS) for at least 3 months, in whom treatment of only one upper limb is necessary for the duration of the study;
* 2b. [Canada] Participants with stable post-stroke ULS for at least 3 months, in whom treatment of only one upper limb is necessary for the duration of the study
* Participants who are either naïve to Botulinum toxin type A (BoNT-A) for ULS or who have been previously treated with BoNT-A for ULS;
* Participants with MAS score of at least 2 at two muscle groups (one of these two muscles groups should be the PTMG) and at least 1 in the remaining muscle group.
* Participants with DAS score of at least 2 on the Principal Target of Treatment (PTT) (one of four functional domains: dressing, hygiene, limb position and pain);
* Participants who require BoNT-A injection in all of the following muscles: flexor carpi radialis, flexor carpi ulnaris, flexor digitorum profundus, flexor digitorum superficialis and biceps brachii;
* Participants for whom injection of a total dose of 900 Units aboBoNT-A or 360 Units onaBoNT-A is considered by the investigator to be clinically appropriate;
* Participants who have been stable for at least 3 months prior to study entry in terms of oral antispasticity, anticoagulant and/or anticholinergic medication if treated are considered by the investigator likely to remain stable for the duration of the study;

Exclusion Criteria:

* Major limitations in the passive range of motion in the paretic upper limb;
* Major neurological impairment (other than limb paresis) that could negatively affect functional performance;
* Participants clinically requiring injection into any upper limb muscles other than the five muscles of one arm listed in Section 5.1, or requiring injection into both arms or any lower limb within the timeframe of the study;
* Hypersensitivity to any BoNT product or excipients;
* Hypersensitivity to cow's milk protein (casein);
* Infection at the proposed injection site(s);
* Known peripheral motor neuropathic diseases, amyotrophic lateral sclerosis or neuromuscular junction disorders (e.g. myasthenia gravis or Lambert-Eaton syndrome);
* Any medical condition (including dysphagia or breathing difficulties/compromised respiratory function) that in the opinion of the investigator, might jeopardize the participant's safety;
* Women who are pregnant or lactating
* Participants treated with BoNT of any type for any indication (e.g. bladder injection, headache or cosmetic) within the previous 12 weeks or planned/likely to be treated during the course of the study;
* Prior history of non-responsiveness to BoNT treatment;
* Previous surgery, or administration of alcohol or phenol in the study limb 6 months or earlier from study enrolment or planned/likely to be treated during the course of the study;
* Participants treated with intrathecal baclofen (except if treatment has reached a stable dose for >4 weeks and is likely to remain stable throughout the study), aminoglycosides or other agents interfering with neuromuscular transmission (e.g. curare-like agents) within the 4 weeks prior to study enrolment or planned/likely to be treated during the course of the study
* BoNT naïve participants with a history of facial neurogenic disorder (facial paralysis, polyradiculoneuropathy) (only for France).
* Participants receiving concomitant medication treatment with the following PT/OT interventions on the study limb: new splinting/orthotics/casting, serial casting, shockwave therapy, dry needling and needle tenotomies. However, PT/OT interventions not intended to reduce study limb spasticity (e.g. functional training exercises) or with a transient (<1 day) reduction of study limb spasticity (e.g. stretching, weight bearing) are allowed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment-emergent Adverse Events (TEAEs) | from baseline (injection) to 12 weeks (injection cycle 1 and 2, each cycle is a maximum 24 weeks))

SECONDARY OUTCOMES:
Rate of Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) | from baseline (injection) to 12 weeks (injection cycle 1 and 2, each cycle is a maximum 24 weeks))
Duration of response | baseline (injection) to retreatment criteria met, from week 10 up to week 24 (for each cycle, 1&2) or baseline to withdrawal or end of study if retreatment criteria not met, up to 24 weeks (for each cycle,1&2, each cycle is a maximum 24 weeks)
Muscle tone assessed by Modified Ashworth scale (MAS) total score | at baseline (injection), 1 week, 4 weeks, 10 weeks, 12 weeks and additional visits at 16 weeks, 20 weeks, 24 weeks (injection cycle 1 and 2; each cycle is a maximum 24 weeks)
  MAS is a scale which represents improvement in spasticity. This tool assesses muscle tone using a six-point scale from 0 = no change to 4 = considerable increase of affected/rigid region.
Perceived function and pain assessed by the Disability Assessment Scale (DAS) total score | at baseline (injection), 1 week, 4 weeks, 10 weeks, 12 weeks and additional visits at 16 weeks, 20 weeks, 24 weeks (injection cycle 1 and 2; each cycle is a maximum 24 weeks)
  DAS scale to determine the extent of functional impairment in four domains: hygiene, dressing, limb position and pain. Impairment will be assessed on a four-point scale (range 0 to 3, where 0 indicates no disability and 3 indicates severe disability). The four domain ratings will be added to give an overall score between 0 and 12.
Physician global assessment (PGA) of treatment response | at baseline (injection), 1 week, 4 weeks, 10 weeks, 12 weeks and additional visits at 16 weeks, 20 weeks, 24 weeks (injection cycle 1 and 2; each cycle is a maximum 24 weeks)
  PGA answers will be made on a nine-point rating scale (from -4 = markedly worse, to +4 = markedly improved).
Change in Quality of Life (QoL) using the SF-12 perceived health score | at baseline (injection), 4 weeks, 12 weeks and at end of each cycle (injection cycle 1 and 2; each cycle is a maximum 24 weeks)
  12-Item Short-form Health Survey (SF-12) is a health survey that will assess general health and wellbeing. The SF-12 summary score is between 0 and 100, with higher scores indicating better self-reported health.
Change in Quality of Life (QoL) using SQoL-6D | at baseline (injection), 4 weeks, 12 weeks and at end of each cycle (injection cycle 1 and 2; each cycle is a maximum 24 weeks)
  Spasticity-related Quality of Life Tool (SQoL-6D) is a brief questionnaire in six domains (pain/discomfort, involuntary movements or spasms, restricted range of movement, caring for the affected limb, using the affected limb and mobility/balance) using a five-level scale ranging from 0 to 4, with higher scores meaning worse condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (76):
- United States (54):
  - University of Alabama, Birmingham, Alabama
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - The University of Arizona, Tucson, Arizona
  - Rancho Los Amigos National Rehabilitation Center (RLANRC) - Neurology, Downey, California
  - Parkinson's & Movement Disorders Institute, Fountain Valley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Loma Linda University Health Care, Loma Linda, California
  - Southland Neurologic Institute, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - Hasbani And Hasbani Medical Group, New Haven, Connecticut
  - Ki Health Partners LLC D/B/A New England Institute for Clinical Research, Stamford, Connecticut
  - First Choice Neurology, Boca Raton, Florida
  - James A Haley Veterans Hospital, Tampa, Florida
  - University of South Florida Health-Morsani Center for Advanced Healthcare, Tampa, Florida
  - Emory University of School of Medicine, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Shirley Ryan Ability Lab, Chicago, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Kansas City Bone and Joint Clinic, P.A. (KCBJ) - Overland Pa, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - LSU Healthcare network, New Orleans, Louisiana
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - William Beaumont Hospital, Dearborn, Michigan
  - Medical Rehabilitation Group, PC, Grand Blanc, Michigan
  - Mary Free Bed Rehabilitation Hospital, Grand Rapids, Michigan
  - Beaumont Hospital, Grosse Pointe, Grosse Pointe, Michigan
  - Michigan Center of Medical Research, Grosse Pointe, Michigan
  - Rusk Rehabilitation Center, Columbia, Missouri
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Cooper University Health Care, Cherry Hill, New Jersey
  - New York University, New York, New York
  - Weill Cornell Medicine Clinical and Translational Science Center, New York, New York
  - North Suffolk Neurology, Port Jefferson, New York
  - Mayo Clinic, Rochester, New York
  - Sunnyview Rehabilitation Hospital, Schenectady, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic - Neurological Institute, Cleveland, Ohio
  - MossRehab - Einstein Medical Center, Elkins Park, Pennsylvania
  - Penn State Health Physical Medicine and Rehabilitation - Neurology, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Aether Medicine, Wayne, Pennsylvania
  - Siskin Hospital for Rehabilitation - Neurology, Chattanooga, Tennessee
  - The Vanderbilt Clinic, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - TIRR Memorial Hermann Research Center, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Carilion Clinic Institute of Orthopaedics and Neurosciences, Roanoke, Virginia
  - MedStar National Rehabilitation Network, Columbia, Washington
  - Swedish Neuroscience Institute, Seattle, Washington
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (4):
  - Lawson Health Research Institute, London, Ontario
  - Moncton Hospital, Moncton
  - Genge Partners, Montreal
  - Victoria General Hospital, Victoria
- France (17):
  - Centre Les Capucins, Angers
  - Hôpital Pellegrin CHU Bordeaux, Bordeaux
  - Hopital Sud, Échirolles
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - Hôpital Saint-Jacques (CHU Nantes), Nantes
  - Hopital Archet (CHU de Nice), Nice
  - Hopital Fernand Widal, Paris
  - Centre Mutualiste de Rééducation et de Réadaptation Fonction, Ploemeur
  - Hôpital Jean Bernard (CHU Poitiers), Poitiers
  - Hôpital Pontchaillou (CHU Rennes), Rennes
  - Pole Saint Helier, Rennes
  - Centre de Perharidy, Roscoff
  - Centre Hospitalier de Saint-Amand-les-Eaux, Saint-Amand-les-Eaux
  - Centre Hospitalier de Saint Amand Montrond, Saint-Amand-Montrond
  - Hopital Henry Gabrielle (HCL), Saint-Genis-Laval
  - Hopitaux Universitaires De Strasbourg, Strasbourg
  - Hopital de Rangueil, Toulouse
- University of Puerto Rico, Santurce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Esquenazi A, Ayyoub Z, Verduzco-Gutierrez M, Maisonobe P, Otto J, Patel AT. AbobotulinumtoxinA Versus OnabotulinumtoxinA in Adults with Upper Limb Spasticity: A Randomized, Double-Blind, Crossover Study Protocol. Adv Ther. 2021 Nov;38(11):5623-5633. doi: 10.1007/s12325-021-01896-3. Epub 2021 Sep 25. PMID 34562231